CLINICAL TRIAL: NCT06536140
Title: The Lived Experiences of Persons With Early Stage Non-small Cell Lung Cancer and Their Significant Other(s) Following Surgery: a Rapid Ethnographic Approach
Acronym: LEILA
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Chris Burtin, Associate Professor, Hasselt University
Other Study IDs: Z-2023064
Record Dates: First submitted 2024-02-14; First posted 2024-08-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NSCLC patients 1-3 months after lung resection surgery with or without (neo-)adjuvant therapy: This study will include twenty persons who underwent surgery for early stage I-IIIA NSCLC (with or without (neo-) adjuvant chemotherapy/radiotherapy/immunotherapy) one to three months before inclusion and their carers significant other(s). This can be one person or multiple persons (e.g. partner, parent, child, brother, sister).
  Interventions: Other: Home observations and interview

INTERVENTIONS:
Other: Home observations and interview — If persons want to participate, the person will be invited one week before the first observation for a 'warm-up' phone call (W1) as a preparation for the three observations and follow-up interview.
  During the observations, SH will be an active participant, offering to help with activities of daily life with the person, so opportunities are created to observe and ask questions (sensory ethnography). The person will be asked to take pictures or make drawings of important things in the house as the observer will be able to better understand how they feel about exercise and PA (visual ethnography). Six weeks after the last observation (W10), formal follow-up interviews (30-60 min) with questions based on the observations that took place, will be held to explore specific issues in-depth.

SUMMARY:
To understand the lived experiences, thoughts and habits about exercise and PA of persons with early stage non-small cell lung cancer and their significant other(s) following surgery.

DETAILED DESCRIPTION:
It is important to gather information on the lived lives of persons and their significant other(s) following surgery for early stage non-small cell lung cancer (NSCLC). The adaptations these persons make, the challenges they face and their personal experiences need to be investigated so their thoughts and habits about exercise and physical activity (PA) can be better understood. In this way, rehabilitation programs focused on exercise and PA can be better individualized. The individualization of such programs is heavily influenced by the person's experiences, including beliefs and expectations regarding exercise and PA. Observations of and informal conversations with persons with early stage NSCLC and their significant other(s) following surgery will offer insight into the challenges faced by these individuals and the opportunities for exercise and PA, how this does and could fit, within their everyday lives so this can be enhanced. It is important to align exercise and PA to everyday activities, to make it meaningful to individuals (more likely to engage) and to obtain sustained effects in the long term. The investigators expect this study to show the highly personal views and behaviour of these persons, warranting an equally personal communication approach to discuss these issues with these persons in light of developing individualized rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Persons who got surgery for early stage I-IIIA NSCLC, one to three months before inclusion;
* If persons received adjuvant chemotherapy/radiotherapy, the inclusion window is one to three months after the end of adjuvant chemotherapy/radiotherapy. If persons receive adjuvant immunotherapy after the end of adjuvant chemotherapy, persons can be included during the immunotherapy;
* Adults (18+ year);
* Ability to give informed consent.

Exclusion Criteria:

* Persons having progressive or recurrent lung cancer;
* Persons who had other malignancies in the last 2 years;
* Persons who do systematically perform or plan to perform structured exercise;
* Persons not living independently at home (e.g. care home, psychiatric institution);
* Psychiatric or cognitive disorders;
* Not understanding and speaking Dutch;
* Not living at home (e.g. nursing home, prison …).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include twenty persons who underwent surgery for early stage I-IIIA NSCLC (with or without (neo-) adjuvant chemotherapy/radiotherapy/immunotherapy) one to three months before inclusion and their carers significant other(s). This can be one person or multiple persons (e.g. partner, parent, child, brother, sister). In case the person doesn't have a significant other, this person will not be excluded from the study. Purposive sampling will be applied. The study will aim to recruit persons with a wide range of characteristics including age, sex and ethnic cultural background as it is important to recruit a diverse sample. We will not have access to the socio-economic background of persons during the screening process.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Barriers and facilitators for exercise and physical activity | Visit 1 during week 1
  Self-developed questionnaire to assess person's motivation and self-efficacy regarding exercise and PA based on Chan et al. (2022) and Rogers et al. (2006)
Motivation and self-efficacy | Visit 1 during week 1
  Exercise Self-Efficacy Scale (ESES), Tampa Scale for Kinesiophobia (TSK), Perceived physical activity questionnaire (LIVAS), SRQ-E (Exercise self-regulation questionnaire)

SECONDARY OUTCOMES:
Socio-demographic information | Visit 1 during week 1
  Name, birth date, address, telephone number, smoking status
Anthropometric information | Visit 1 during week 1
  Weight in kg, height in cm
Medical history (from medical file) | Before visit 1
  Oncological history, pathological staging (TNM 8e edition), treatment type, medication, hospital admissions in the past year
Lung function (from medical file) | Before visit 1
  Complete lung function after surgery
Physical activity | One week between the third week and fourth week.
  Objectively measured physical activity: Mean steps per day, MVPA, daily walking time, movement intensity during walking, sedentary time (measured by Dynaport MoveMonitor and Actigraph)
Activity related information | Visit 2 during week 2
  Previous exercise/activity interventions. Marital status, living status, education level, last work experience, current work status, feeling of loneliness, having grandchildren and/or a pet(s), experience with step counters/activity trackers
Comorbidities | Visit 2 during week 2
  Self-Administered Comorbidity Questionnaire
Symptoms of dyspnea | Visit 2 during week 2
  Modified Medical Research Council Dyspnoe vragenlijst (mMRC)
Symptoms of fatigue | Visit 2 during week 2
  Multidimensional Fatigue Inventory (MFI-20)
Symptoms of anxiety | Visit 3 during week 3
  Depression Anxiety Stress Scale (DASS-21)
Health related Quality of Life | Visit 3 during week 3
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30), European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire and Lung Cancer Module (EORTC QLQ-LC-13) and EuroQoL five-dimensional instrument (EQ-5D)
Quality of Life | Visit 3 during week 3
  36-Item Short Form Survey (SF-36) and 12-Item Short Form Survey (SF-12)
Loneliness | Visit 3 during week 3
  Loneliness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Chris Burtin, PhD, Principal Investigator — University Hasselt
Locations (1):
- Faculteit Revalidatiewetenschappen - Gebouw 7, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No